CLINICAL TRIAL: NCT00673153
Title: Phase II Trial of Vorinostat (Suberoylanilide Hydroxamic Acid or SAHA; Zolinza™) in Combination With Gemtuzumab Ozogamicin (Mylotarg™) as Induction and Post-Remission Therapy in Older Patients With Previously Untreated Non-M3 Acute Myeloid Leukemia
Brief Title: Vorinostat and Gemtuzumab Ozogamicin in Treating Older Patients With Previously Untreated Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roland Walter, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2200.00; NCI-2010-00401 (Registry Identifier: National Cancer Institute (NCI))
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Gemtuzumab; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): REMISSION INDUCTION THERAPY: Patients receive oral vorinostat once daily on days 1-9 and gemtuzumab ozogamicin IV over 2 hours on day 8. Treatment repeats every 15-22 days for up to 3 courses. .
  CONSOLIDATION THERAPY: Beginning within 60 days after the completion of remission induction therapy, patients receive oral vorinostat once daily on days 1-9 and gemtuzumab ozogamicin IV over 2 hours on day 8.
  MAINTENANCE THERAPY: Patients receive oral vorinostat once daily on days 1-14. Treatment repeats every 28 days for 4 courses.
  Interventions: Drug: gemtuzumab ozogamicin; Drug: vorinostat; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gemtuzumab ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; hP67.6-Calicheamicin; Mylotarg; WAY-CMA-676
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: Vorinostat may stop the growth of cancer cells by interfering with various proteins needed for cell growth. Monoclonal antibodies, such as gemtuzumab ozogamicin (GO), can block cancer growth in different ways. GO finds cancer cells and helps kill them by carrying a cancer-killing substance to them. Giving vorinostat together with gemtuzumab ozogamicin may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving vorinostat together with gemtuzumab ozogamicin works in treating older patients with previously untreated acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the CR/CRi rate after treatment with vorinostat plus GO. (Good risk group) II. To determine the 30-day survival after treatment with vorinostat plus GO. (Poor risk group)

SECONDARY OBJECTIVES:

I. To estimate the frequency and severity of regimen-associated toxicities, along with 30-day survival after start of treatment with vorinostat plus GO. (Good risk group) II. To determine the CR/CRi rate after treatment with vorinostat plus GO, and estimate the frequency and severity of regimen-associated toxicities. (Poor risk group) III. To investigate the relapse-free survival of patients who achieve CR/CRi and receive maintenance therapy on this study.

IV. To define cellular factors associated with clinical response to GO/vorinostat and determine the mechanisms underlying the synergistic effect between GO and vorinostat on primary AML cells (in vitro correlative and mechanistic studies).

OUTLINE:

REMISSION INDUCTION THERAPY: Patients receive oral vorinostat once daily on days 1-9 and gemtuzumab ozogamicin IV over 2 hours on day 8. Treatment repeats every 15-22 days for up to 3 courses.

CONSOLIDATION THERAPY: Beginning within 60 days after the completion of remission induction therapy, patients receive oral vorinostat once daily on days 1-9 and gemtuzumab ozogamicin IV over 2 hours on day 8.

MAINTENANCE THERAPY: Patients receive oral vorinostat once daily on days 1-14. Treatment repeats every 28 days for 4 courses.

All treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Morphological diagnosis of AML other then acute promyelocytic leukemia (FAB M3) according to WHO diagnostic criteria; diagnosis of AML must be based on bone marrow or peripheral blood studies obtained within 28 days prior to study registration or start of hydroxyurea (for patients presenting with WBC >= 10,000/uL), and no potentially anti-leukemic therapy (with the exception of hydroxyurea) must have been given between AML diagnosis and study registration; a bone marrow biopsy is not routinely required but should be obtained if the aspirate is dilute, hypocellular, or inaspirable; outside bone marrows performed within the stipulated time period are acceptable as long as the slides are reviewed at a study institution
* Cytogenetic analysis on bone marrow or peripheral blood specimen is available; based on the result from the first interim analysis, patients stratified into the good-risk group are only eligible if their AML has favorable cytogenetics (core-binding factor AML) or has a normal karyotype; patients stratified into the poor-risk group are eligible independent of the cytogenetic analysis
* Pretreatment bone marrow and peripheral blood specimens for correlative studies are available; if bone marrow was performed at an outside facility, submission of peripheral blood only is acceptable as long as the peripheral blast count is > 5,000/uL and > 50% of total WBC
* Patients with a history of antecedent MDS are eligible, if prior treatment did not include intensive chemotherapy; patients may have received hematopoietic growth factors, thalidomide/lenalidomide, 5-azacytidine/decitabine, arsenic trioxide, signal transduction inhibitors, or low dose cytarabine (< 100 mg/m2/day) for treatment of MDS; patients must be off prior therapy for MDS at least 30 days prior to study registration, and all non-hematologic toxicities must have resolved to < grade 2
* ECOG/WHO/Zubrod performance status of 0-3
* Bilirubin =< 2.5 x Institutional Upper Limit of Normal (IULN) unless elevation is thought to be due to hepatic infiltration by AML, Gilbert's syndrome, or hemolysis (assessed within 14 days prior to registration)
* SGOT (AST) and SPGT (ALT) =< 1.5 x IULN unless elevation is thought to be due to hepatic infiltration by AML (assessed within 14 days prior to registration)
* Serum creatinine =< 1.5 x IULN (assessed within 14 days prior to registration)
* Left ventricular ejection fraction >= 40% and no clinical evidence of congestive heart failure (assessed within 28 days prior to registration, e.g. by MUGA scan or echocardiography)
* Men of reproductive potential must use an effective contraceptive method throughout the study and for a period of at least 3 months after the study
* Women must be postmenopausal; a postmenopausal woman is defined as a woman who has experienced amenorrhea > 12 consecutive months or a woman on hormone replacement therapy with documented FSH level > 35 mIU/mL (women of childbearing potential must have a pregnancy test within 28 days prior to registration, and must use an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 3 months after the study)
* Provide signed written informed consent
* Willingness to undergo bone marrow examination on day 8 of first induction cycle
* WBC < 10,000/uL (patients with WBC >= 10,000/uL must undergo cytoreduction with hydroxyurea prior to enrollment and will not be enrolled if the WBC remains >= 10,000/uL (of note, patients with symptoms/signs of hyperleukocytosis or WBC > 100,000/uL can be treated with leukapheresis prior to enrollment)

Exclusion Criteria:

* Diagnosis of another malignancy, unless the patient was diagnosed at least 2 years earlier and has been disease-free for at least 6 months following the completion of curative intent therapy; there should be no plan to begin therapy for the prior malignancy at the time of study registration; prior treatment with AML induction-type chemotherapy is not allowed (note the following exceptions: patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed; patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen [PSA] values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed; concurrent hormonal therapy is allowed)
* Myeloid blast crisis of chronic myelogenous leukemia (CML)
* Prior systemic chemotherapy for AML with the exception of hydroxyurea
* Prior treatment with AML induction-type chemotherapy, GO, HDAC inhibitors, or high dose chemotherapy with hematopoietic stem cell support
* Treatment with HDAC inhibitors during the last 3 years prior to registration, including the use of valproic acid for seizure activity or other purposes
* Known hypersensitivity to hydroxyurea, GO, or vorinostat
* Clinical evidence suggestive of central nervous system (CNS) involvement with leukemia unless a lumbar puncture confirms the absence of leukemic blasts in the cerebrospinal fluid (CSF)
* Prior positive test for the human immunodeficiency virus (HIV)
* Breastfeeding
* Uncontrolled systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-03; Primary Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Walter, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walter RB, Medeiros BC, Powell BL, Schiffer CA, Appelbaum FR, Estey EH. Phase II trial of vorinostat and gemtuzumab ozogamicin as induction and post-remission therapy in older adults with previously untreated acute myeloid leukemia. Haematologica. 2012 May;97(5):739-42. doi: 10.3324/haematol.2011.055822. Epub 2011 Dec 1. PMID 22133771

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: REMISSION INDUCTION THERAPY: Patients receive oral vorinostat once daily on days 1-9 and gemtuzumab ozogamicin IV over 2 hours on day 8. Treatment repeats every 15-22 days for up to 3 courses. .
  CONSOLIDATION THERAPY: Beginning within 60 days after the completion of remission induction therapy, patients receive oral vorinostat once daily on days 1-9 and gemtuzumab ozogamicin IV over 2 hours on day 8.
  MAINTENANCE THERAPY: Patients receive oral vorinostat once daily on days 1-14. Treatment repeats every 28 days for 4 courses.
  gemtuzumab ozogamicin: Given IV
  vorinostat: Given orally
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Arm I
Started | 31
Completed | 30
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 31
Age, Continuous [Mean (Full Range); unit: years] | 72 [61 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 31
Risk Group [Count of Participants; unit: Participants] — Poor-risk Group: patients aged ≥70 years and performance status 2-3; Good-risk Group: aged 60-69 years with performance status 0-3, or aged ≥70 years and performance status 0-1
  Performance status based on Eastern Cooperative Oncology Group's scale, abbreviated below:
  0 Fully active
  1. Restricted in strenuous activity but capable of a light or sedentary work activities,
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities;
  3. Capable of only limited selfcare;
  4. Completely disabled; cannot carry on any selfcare; confined to bed or chair
  5. Dead
  Participants
    Poor-risk Group | 10
    Good-risk Group | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving CR or CRi With Induction Therapy (Good-risk Group)
Time Frame: after completion of induction therapy, administered every 21-42 days for up to two courses
Population: Good-risk Group: aged 60-69 years with performance status 0-3, or aged ≥70 years and performance status 0-1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 21
Participants | 6

2. Primary Outcome: Number of Participants Alive at Day 30 (Poor-risk Group)
Time Frame: At day 30
Population: Poor-risk Group: patients aged ≥70 years and performance status 2-3
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 10
Participants | 8

3. Secondary Outcome: Relapse-free Survival (Good- and Poor-risk Group)
Time Frame: At relapse
Population: Poor-risk Group: patients aged ≥70 years and performance status 2-3; Good-risk Group: aged 60-69 years with performance status 0-3, or aged ≥70 years and performance status 0-1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 31
Participants | 7

4. Secondary Outcome: Number of Participants Achieving CR or CRi With Induction Therapy (Poor-risk Group)
Time Frame: after completion of induction therapy, administered every 21-42 days for up to two courses
Population: Poor-risk Group: patients aged ≥70 years and performance status 2-3
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 10
Participants | 1

5. Secondary Outcome: Number of Participants Alive at Day 30 (Good-risk Group)
Time Frame: At day 30
Population: Good-risk Group: aged 60-69 years with performance status 0-3, or aged ≥70 years and performance status 0-1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 21
Participants | 20

ADVERSE EVENTS:
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 12/31
Other Adverse Events (participants affected / at risk) | 29/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=31)
GI Bleed (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Death (General disorders) | 4 (4)
Neutropenic Fever (Infections and infestations) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Bleeding at PICC site (Surgical and medical procedures) | 1 (1)
Perirectal cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 1 (1)
E-coli Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=31)
Neutropenia (Blood and lymphatic system disorders) | 19 (26)
Neutropenic Fever (Infections and infestations) | 7 (14)
Thrombocytopenia (Blood and lymphatic system disorders) | 18 (22)
Anemia (Blood and lymphatic system disorders) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chills (General disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Edema/Swelling (General disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Headache (Nervous system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Weight loss (Investigations) | 2 (2)
Chest pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Gingival bleeding (Gastrointestinal disorders) | 1 (2)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Confusion (Psychiatric disorders) | 2 (2)
Creatinine increased (Investigations) | 3 (3)
Blurred Vision (Eye disorders) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
White blood cell decreased (Blood and lymphatic system disorders) | 2 (3)
Pulmonary Nodules (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Increased urinary frequency (Renal and urinary disorders) | 1 (1)
Diaphoresis (Metabolism and nutrition disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Increased lactate dehydrogenase (Investigations) | 1 (1)
Malaise (General disorders) | 1 (1)
Hematoma, scalp (Vascular disorders) | 1 (1)
Gastrointestinal Bleed (Gastrointestinal disorders) | 2 (2)
Appendix Fistula (Gastrointestinal disorders) | 1 (1)
Hemorrhage, post bone marrow (Blood and lymphatic system disorders) | 1 (1)
Streptococcus salivarius (Immune system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Bacteremia (Infections and infestations) | 3 (3)
Cardiac arrhythmia (Cardiac disorders) | 2 (5)
Heart Failure (Cardiac disorders) | 1 (2)
Orthostatic hypotension (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Non-ST-elevation myocardial infarction (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor CAN require changes to the communication and CAN extend the embargo.